CLINICAL TRIAL: NCT00412451
Title: A Randomized, Sham-Injection Controlled, Double-Masked, Ascending-Dose, Dose-Range-Finding Trial of Microplasmin Intravitreal Injection for Non-Surgical Posterior Vitreous Detachment (PVD) Induction for Treatment of DME.
Brief Title: A Multicenter Study to Compare Multiple Doses of Intravitreal Microplasmin Versus Sham Injection for Treatment of Patients With Diabetic Macular Edema (DME)
Acronym: MIVI-II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ThromboGenics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TG-MV-002
Record Dates: First submitted 2006-12-14; First posted 2006-12-18 (Estimated); Results first posted 2013-09-13 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-04

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; PVD; DME; Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — microplasmin; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ocriplasmin 25µg (Experimental): 25µg ocriplasmin intravitreal injection versus sham injection
  Interventions: Drug: ocriplasmin
- Ocriplasmin 75µg (Experimental): 75µg ocriplasmin intravitreal injection versus sham injection
  Interventions: Drug: ocriplasmin
- Ocriplasmin 125µg (Experimental): 125µg ocriplasmin intravitreal injection versus sham injection
  Interventions: Drug: ocriplasmin
- sham injection (Sham Comparator): Sham injection
  Interventions: Other: Sham injection

INTERVENTIONS:
Drug: ocriplasmin — Intravitreal injection, single administration
  Other Names: microplasmin
  Arms: Ocriplasmin 125µg; Ocriplasmin 25µg; Ocriplasmin 75µg
Other: Sham injection — Sham intravitreal injection
  Arms: sham injection

SUMMARY:
A multicenter study to compare multiple doses of intravitreal microplasmin for non-surgical PVD induction for treatment of patients with DME.

ELIGIBILITY:
Inclusion Criteria include:

* patients >18 years of age with Diabetic Macular Edema

Exclusion Criteria include:

* PVD present at baseline
* Vitreous hemorrhage
* Certain vitreoretinal conditions including proliferative disease, rhegmatogenous retinal detachment, and proliferative vitreoretinopathy (PVR)
* Patients who have had a vitrectomy in the study eye at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-12; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- Belgium (3):
  - ZNA OCMW Antwerpen, Antwerp
  - University Hospital of Ghent, Ghent
  - University Hospital Leuven, Leuven
- Ludwig Maximillian University, Munich, Germany
- Italy (4):
  - University of Milan, Milan
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Institute of Ophtalmology, Policlinico A: Gemelli (University Hospital),Catholic University of Sacred Heart, Rome
  - Ospedale di Circolo di Varese, Insubria University, Varese
- Netherlands (2):
  - Academic Hospital Groningen, Groningen
  - Het Oogziekenhuis Rotterdam, Rotterdam
- Spain (3):
  - Institut de Microcirurgia Ocular de Barcelona, Barcelona
  - Hospital Vall D'Hebron, Barcelona
  - Instituto Technologico de Oftalmologia SL., Santiago de Compostela
- United Kingdom (2):
  - Royal Liverpool & Broadgreen Hospital, Liverpool
  - Moorfields Eye Hospital, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled on 15 December 2006 and the last patient completed the last visit on 19 January 2010. All patients were selected in medical clinics
Pre-assignment Details: The trial investigated 3 doses: 25, 75 and 125µg in 3 consecutive cohorts. Patients in each cohort were to be randomized to active treatment or sham injection in a 3:1 ratio. Enrolment into the high dose microplasmin groups was to start only after acceptable safety had been achieved with the previous doses as determined by a Study Safety Committee.
Groups:
- Ocriplasmin 25µg: 25µg ocriplasmin intravitreal injections versus sham injection
- 0criplasmin 125µg: 125µg ocriplasmin intravitreal injection versus sham injection
Period: Overall Study
Arm/Group | Ocriplasmin 25µg | Ocriplasmin 75µg | 0criplasmin 125µg | Sham Injection
Started | 8 | 15 | 15 | 13
Completed | 8 | 15 | 14 | 11
Not Completed | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Sham Injection: Sham injection
  Sham injection : Sham intravitreal injection
- Total: Total of all reporting groups
Arm/Group | Ocriplasmin 25µg | Ocriplasmin 75µg | Ocriplasmin 125µg | Sham Injection | Total
Number analyzed (Participants) | 8 | 15 | 15 | 13 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (9.8) | 67.3 (8.8) | 61.7 (13.4) | 69.9 (6.2) | 63.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 4 | 4 | 19
  Male | 3 | 9 | 11 | 9 | 32

OUTCOME MEASURES:

1. Primary Outcome: PVD Induction
Description: The primary efficacy variable was the proportion of patients with total posterior vitreous detachment (PVD) on Day 14 as determined by a masked central reading center (CRC) using 4-quadrant B-scan and optical coherence tomography (OCT)
Time Frame: Day 14 post-injection
Population: Intent-To-Treat (ITT), Last Observation Carried Forward (LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Ocriplasmin 25µg | Ocriplasmin 75µg | Ocriplasmin 125µg | Sham Injection
Number analyzed (Participants) | 8 | 15 | 15 | 13
percentage of participants | 0 | 20 | 13.3 | 30.8
Statistical Analysis 1: Comparison: Ocriplasmin 25µg vs Sham Injection; Test type: Superiority or Other; p = 0.131, Fisher Exact; Odds Ratio (OR) = 0.001, 95% CI 2-sided [0.001 to 999.999]
Statistical Analysis 2: Comparison: Ocriplasmin 75µg vs Sham Injection; Test type: Superiority or Other; p = 0.670, Fisher Exact; Odds Ratio (OR) = 0.562, 95% CI 2-sided [0.132 to 2.400]
Statistical Analysis 3: Comparison: Ocriplasmin 125µg vs Sham Injection; Test type: Superiority or Other; p = 0.372, Fisher Exact; Odds Ratio (OR) = 0.346, 95% CI [0.070 to 1.703]

ADVERSE EVENTS:
Time Frame: AEs/SAEs were collected from injection day up to Month 12 post-injection
Arm/Group | Ocriplasmin 25µg | Ocriplasmin 75µg | Ocriplasmin 125µg | Sham Injection
Serious Adverse Events (participants affected / at risk) | 1/8 | 4/15 | 5/15 | 9/13
Other Adverse Events (participants affected / at risk) | 1/8 | 4/15 | 5/15 | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocriplasmin 25µg (N=8) | Ocriplasmin 75µg (N=15) | Ocriplasmin 125µg (N=15) | Sham Injection (N=13)
maculopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infaction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Optic disc vascular disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Monoparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ocriplasmin 25µg (N=8) | Ocriplasmin 75µg (N=15) | Ocriplasmin 125µg (N=15) | Sham Injection (N=13)
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
Maculopathy (Eye disorders) | 0 | 0 | 0 | 1
Macular oedema (Eye disorders) | 0 | 1 | 0 | 0
Optic disc vascular disorder (Eye disorders) | 0 | 1 | 0 | 0
Retinal artery occlusion (Eye disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1
Monoparesis (Nervous system disorders) | 0 | 0 | 1 | 0
Heamatoma (Vascular disorders) | 0 | 0 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less